CLINICAL TRIAL: NCT00092508
Title: Phase 3, Multi-Center, Randomized, Double-Blind, Parallel-Arm, 52-Week Dose Comparison Study of the Efficacy and Safety of 25 mg QD and 50 mg QD of OPC-6335 Oral Tablets and 800 mg BID of Asacol® in the Maintenance of Ulcerative Colitis Remission
Brief Title: CORE: A Study of OPC-6535 With Asacol® in Maintaining Ulcerative Colitis (UC) Remission
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 197-02-220
Record Dates: First submitted 2004-09-22; First posted 2004-09-28 (Estimated); Last update posted 2007-06-21 (Estimated); Status verified 2007-06

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis Remission; ulcerative; colitis; remission; relapse; Asacol®; maintain; maintenance; flare; rectal; bleeding; bowel
MeSH Terms: conditions — Colitis, Ulcerative; Ulcer; Colitis; Recurrence; Hemorrhage | interventions — tetomilast; Mesalamine

INTERVENTIONS:
Drug: OPC-6535
Drug: Asacol®

SUMMARY:
This dose comparison study, taking place at over 200 sites worldwide, will compare the dosing, safety and efficacy of an investigational medicine OPC-6535 to the dosing, safety and efficacy of Asacol ® in the maintenance of remission in subjects with ulcerative colitis.

DETAILED DESCRIPTION:
Objective(s):

This study will compare the safety and efficacy of 25 mg per day (QD) and 50 mg QD of OPC-6535 to 800 mg twice a day (BID) of Asacol® in the maintenance of remission in subjects with ulcerative colitis.

Subject Population:

* Subjects with ulcerative colitis currently in remission defined as rectal bleeding (RB) and flexible sigmoidoscopy (FS) scores of 0, on or off a stable dose of sulfasalazine or 5-ASA products for at least 6 weeks.
* Subjects must have had the diagnosis of ulcerative colitis established by prior colonoscopy or undergo colonoscopy in lieu of flexible sigmoidoscopy during the Screening Period.
* Subjects must have had treatment for a flare of ulcerative colitis, with symptomatic onset of remission occurring no more than 52 weeks from the Screening Period.
* Subjects may not have used corticosteroids, topical agents (corticosteroid or 5-ASA enemas, suppositories, foams), azathioprine, 6-mercaptopurine, or methotrexate within 6 weeks of the Screening Period. Upon entry, sulfasalazine and 5-ASA containing products will be discontinued.

Safety: Vital signs, ECGs, laboratory studies (including hematology, clinical chemistry, and urinalysis), and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18 to 80 years of age, inclusive.
* Subjects with a prior diagnosis of ulcerative colitis, established by colonoscopy.
* Subjects currently in remission.
* Subjects who have undergone treatment for a flare of ulcerative colitis, with symptomatic onset of remission occurring no more than 52 weeks from the Screening Period.
* If subjects are taking sulfasalazine or 5-ASA products prior to entry, the dose must be stable for at least 6 weeks prior to the Screening Period. NOTE: During the study, use of these drugs will be discontinued.
* Subjects having undergone colonoscopy with pan-colonic surveillance biopsies negative for dysplasia within 1 year of the Screening Visit if at increased risk of colorectal cancer (≥ 8 year history of ulcerative colitis).
* Female or male subjects who are surgically sterilized or who are prepared to and agree to practice a double-barrier form of birth control from the Screening Period through 30 days (females) and 90 days (males), respectively, from the last dose of study medication. Females who are more than 12 months post-menopausal are also eligible to participate in the study.

Exclusion Criteria:

* Subjects who have active disease.
* Subjects who have any other clinically significant disease(s) or condition/procedure(s).
* Subjects who have had major gastrointestinal surgery including, but not limited to, a colostomy, an ileostomy or previous colonic surgery other than appendectomy.
* Subjects who have used corticosteroids or topical agents (corticosteroid or 5-ASA enemas, suppositories, foams) within 6 weeks of the Screening Period.
* Female subjects who are pregnant or lactating.
* Other exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1725 (Estimated)
Dates: Start 2004-05; Study Completion 2007-05

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Clinical Research Associates, Huntsville, Alabama
  - West Gastroenterology Medical Group, Los Angeles, California
  - Mark Lamet, Hollywood, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - Advanced Gastroenterology Associates, Palm Harbor, Florida
  - Florida Medical Clinic, Zephyrhills, Florida
  - Digestive Disorders Associates, Annapolis, Maryland
  - Metropolitan Gastroenterology Group, Chevy Cha, Maryland
  - Coastal Research Associates, Braintree, Massachusetts
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Digestive Health Specialists, PA, Tupelo, Mississippi
  - Center for Digestive and Liver Diseases, Mexico, Missouri
  - Atlantic Gastroenterology Associates, PA, Egg Harbor, New Jersey
  - Long Island Clinical Research Associates, Great Neck, New York
  - Asheville Gastroenterology Associates, Asheville, North Carolina
  - Charlotte Gastroenterology & Hepatology, Charlotte, North Carolina
  - Bethany Medical Center, High Point, North Carolina
  - Hanover Medical Specialists, PA, Wilmington, North Carolina
  - GI & Liver Consultants, Dayton, Ohio
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Healthcare Research Consultants, Tulsa, Oklahoma
  - Medical University of South Carolina, Charleston, South Carolina
  - Gastroenterology Associates, Kingsport, Tennessee
  - Gastroenterology Clinic of San Antonio, San Antonio, Texas
  - Advanced Research Institute, Ogden, Utah
  - McGuire DVAMC, Richmond, Virginia